CLINICAL TRIAL: NCT02512406
Title: Sensory Processing in Tourette Syndrome
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400293
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Tourette Syndrome
Keywords: Tourette Syndrome; Tics
MeSH Terms: conditions — Tourette Syndrome; Tics | interventions — Demography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Tourette Syndrome: Questionnaires including the Sensory Profile or the Adult/Adolescent Sensory profile and Children's Yale-Brown Obsessive Compulsive Scale or Yale Global Tic Severity Scale will be administered. When time permits, the Children's Yale-Brown Obsessive Compulsive Scale or Yale-Brown Obsessive Compulsive Scale will also be administered. Demographic data will also be collected for each study patient.
  Interventions: Other: The Sensory Profile; Other: The Adult/Adolescent Sensory Profile; Other: Children's Yale-Brown Obsessive Compulsive Scale; Other: Yale-Brown Obsessive Compulsive Scale; Other: Yale Global Tic Severity Scale; Other: Demographic Data

INTERVENTIONS:
Other: The Sensory Profile — 60 item questionnaire administered to participants age 6-10 with questions pertaining to sensory processing categories of Taste/Smell, Movement, Visual, Touch, Activity Level, and Auditory. Scores are tallied for each category. Results are plotted along an x and y-axis with one axis being perception or stimulus (low registration to sensory sensitivity) and the other being response to stimulus (sensation seeking to sensation avoiding). Each category is plotted along this axis and compared to normative data which is included in this tool.
Other: The Adult/Adolescent Sensory Profile — 60 item questionnaire administered to participants age 11 and older with questions pertaining to sensory processing categories of Taste/Smell, Movement, Visual, Touch, Activity Level, and Auditory. Scores are tallied for each category. Results are plotted along an x and y-axis with one axis being perception or stimulus (low registration to sensory sensitivity) and the other being response to stimulus (sensation seeking to sensation avoiding). Each category is plotted along this axis and compared to normative data which is included in this tool.
Other: Children's Yale-Brown Obsessive Compulsive Scale — 10-item symptom checklist questionnaire administered by a physician to participants aged 6-14. 1st part is a yes/no checklist of obsessions (1-42) and compulsions (43-67) experienced in the past or present. 2nd part is a scored severity scale with 10 questions in which they assign a 0-4 severity score which is summed for a total score.
Other: Yale-Brown Obsessive Compulsive Scale — 10-item symptom checklist questionnaire administered by a physician to participants aged 15 and older. 1st part is a yes/no checklist of obsessions (1-42) and compulsions (43-67) experienced in the past or present. 2nd part is a scored severity scale with 10 questions in which they assign a 0-4 severity score which is summed for a total score.
Other: Yale Global Tic Severity Scale — Clinician administered questionnaire given to all participants. Part 1 asks about 10 types of motor tics, 12 types of vocal tics (current, ever, age of onset, description). Part 2 is a severity rating that scores both motor and vocal tics on a 0-5 scale for each severity item: number of tics, intensity, frequency, complexity, interference, impairment. Totals are summed for all items.
Other: Demographic Data — Data will be collected including: Age, duration of symptoms, presence or absence of autism spectrum disorder, presence or absence of OCD, presence or absence of ADHD.

SUMMARY:
The purpose of this study is to learn more about how patients with Tourette Syndrome deal with sensory stimuli in their environment such as bright lights, loud noises, physical sensations such as shirt tags, etcetera. We will compare responses of patients with Tourette Syndrome to those without Tourette Syndrome.

The study aims to better characterize sensory processing abnormalities by sensory modality: The investigators will use a measuring tool based on Dunn's 1997 model of sensory processing, the Sensory Profile, which will allow the investigator to characterize both registration and response to external stimuli, as well as to delineate which sensory modalities are affected. Identifying which sensory modalities are most affected may guide future research into the pathophysiology of sensory processing abnormalities in TS.

The investigators also aim to correlate sensory processing abnormalities with the presence of Obsessive Compulsive Disorder (OCD), Attention-deficit/hyperactivity disorder (ADHD) , and autism spectrum disorders.

DETAILED DESCRIPTION:
While it is widely recognized that patients with tic and Tourette Syndrome (TS) experience heightened sensitivity to or abnormal processing of internal sensations, it has also been suggested that patients with tic and TS experience abnormal processing of external sensations/stimuli. While this sensitivity to external stimuli does not appear to trigger motor or vocal tics, it can significantly affect quality of life. These sensitivities can be a source of irritation, discomfort, and distraction that can be equally or more disruptive than vocal or motor tics. Heightened sensitivity to external stimuli or other abnormalities of external sensory processing have been identified in other neuropsychological disorders such as autism spectrum disorders, schizophrenia, traumatic brain injury, ADHD, and obsessive-compulsive disorder (OCD) . TS often presents with co-morbid diagnoses including attention-deficit and hyperactivity disorder (ADHD) and obsessive-compulsive disorder (OCD) but it is not currently known whether sensitivity to external stimuli is due to a central processing abnormality common to these disorders.

This study's objective is to use a variety of questionnaires to determine how external stimuli along with the presence of other disorders effect sensory processing.

ELIGIBILITY:
Inclusion Criteria:

* Targeted study population includes patients diagnosed with Tourette Syndrome
* Patient of University of Florida Movement Disorders Center diagnosed with Tourette Syndrome by a movement disorder specialist, according to DSM IV diagnostic criteria
* Age 6-18
* Presence of parent or guardian able to provide consent in the case of minors

Exclusion Criteria:

* Inability of patient or, in the case of minors, parent/guardian to provide informed consent
* Inability of designated person to complete questionnaires. In the case of patients' age 10 and younger, this would refer to the parent/guardian. In the case of patients older than 10, this could be either the patient or their parent/guardian

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Targeted study population includes patients 6-18 diagnosed with Tourette Syndrome who are a patient of University of Florida Movement Disorders Center.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
The Sensory Profile | Day 1
  60 item questionnaire administered to participants age 6-10 with questions pertaining to sensory processing categories of Taste/Smell, Movement, Visual, Touch, Activity Level, and Auditory. Scores are tallied for each category. Results are plotted along an x and y-axis with one axis being perception or stimulus (low registration to sensory sensitivity) and the other being response to stimulus (sensation seeking to sensation avoiding). Each category is plotted along this axis and compared to normative data which is included in this tool.
The Adult/Adolescent Sensory Profile | Day 1
  60 item questionnaire administered to participants age 11 and older with questions pertaining to sensory processing categories of Taste/Smell, Movement, Visual, Touch, Activity Level, and Auditory. Scores are tallied for each category. Results are plotted along an x and y-axis with one axis being perception or stimulus (low registration to sensory sensitivity) and the other being response to stimulus (sensation seeking to sensation avoiding). Each category is plotted along this axis and compared to normative data which is included in this tool.
Children's Yale-Brown Obsessive Compulsive Scale | Day 1
  10-item symptom checklist questionnaire administered by a physician to participants aged 6-14. 1st part is a yes/no checklist of obsessions (1-42) and compulsions (43-67) experienced in the past or present. 2nd part is a scored severity scale with 10 questions in which they assign a 0-4 severity score which is summed for a total score.
Yale-Brown Obsessive Compulsive Scale | Day 1
  10-item symptom checklist questionnaire administered by a physician to participants aged 15 and older. 1st part is a yes/no checklist of obsessions (1-42) and compulsions (43-67) experienced in the past or present. 2nd part is a scored severity scale with 10 questions in which they assign a 0-4 severity score which is summed for a total score.
Yale Global Tic Severity Scale | Day 1
  Clinician administered questionnaire given to all participants. Part 1 asks about 10 types of motor tics, 12 types of vocal tics (current, ever, age of onset, description). Part 2 is a severity rating that scores both motor and vocal tics on a 0-5 scale for each severity item: number of tics, intensity, frequency, complexity, interference, impairment. Totals are summed for all items.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Malaty, M.D., Principal Investigator — University of Florida
Locations (1):
- UF Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States